CLINICAL TRIAL: NCT07007559
Title: ASPEN-09: A Phase 1b/2, Multicenter, Multi Arm Study of Evorpacept in Combination With Anti-cancer Therapies in Advanced / Metastatic Malignancies
Brief Title: ASPEN-09: A Study of Evorpacept in Combination With Anti-cancer Therapies in Advanced / Metastatic Malignancies
Acronym: ASPEN-09
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ALX Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT148009
Record Dates: First submitted 2025-05-22; First posted 2025-06-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer, Metastatic
Keywords: metastatic; Her2+; metastatic HER2-positive breast cancer; breast cancer; HER2-positive; Evorpacept; CD47; ERBB2; Enhertu; trastuzumab deruxtecan; ASPEN-09; Herceptin; solid tumors; trastuzumab; ALX148; mBC; ASPEN-Breast
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — ALX148; Trastuzumab; Paclitaxel; Capecitabine; eribulin; Gemcitabine; Vinorelbine

STUDY DESIGN:
Intervention Model Description: This is a basket study with substudies based on indications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Evorpacept+Trastuzumab+Chemo in participants with metastatic HER2+ breast cancer (Experimental): * Evorpacept (IV) - once every 3 weeks (Q3W)
  * Trastuzumab (IV) - once every 3 weeks (Q3W)
  * Chemotherapy (physician selects one of the following):
    * Capecitabine (Oral) 14 days every 3 weeks
    * Eribulin (IV) twice every 3 weeks
    * Gemcitabine (IV) twice every 3 weeks
    * Paclitaxel (IV) once every 3 weeks (Q3W)
    * Vinolrebine (IV) twice every 3 weeks
  Interventions: Drug: Evorpacept (ALX148); Drug: Trastuzumab; Drug: Paclitaxel; Drug: Capecitabine; Drug: Eribulin; Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Evorpacept (ALX148) — IV infusion
Drug: Trastuzumab — IV infusion
  Other Names: Herceptin
Drug: Paclitaxel — IV infusion
  Other Names: Taxol
Drug: Capecitabine — Oral administration
  Other Names: Xeloda
Drug: Eribulin — IV infusion
  Other Names: Halaven
Drug: Gemcitabine — IV infusion
  Other Names: Gemzar
Drug: Vinorelbine — IV infusion
  Other Names: Navelbine

SUMMARY:
The purpose of this study is to evaluate evorpacept with anti-cancer therapies in advanced/metastatic malignancies. The study is comprised of the following substudies:

* Metastatic HER2+ breast cancer (MBC) - single-arm substudy evaluating the efficacy, safety, and tolerability of evorpacept in combination with trastuzumab and chemotherapy in participants with HER2-positive metastatic breast cancer who have previously received trastuzumab-deruxtecan. This substudy is actively recruiting.
* Metastatic colorectal cancer (CRC) - dose escalation phase to evaluate evorpacept in combination with other drugs. This substudy is not recruiting.
* Recurrent/metastatic head and neck cancer (HNSCC) - dose escalation phase to evaluate evorpacept in combination with other drugs. This substudy is not recruiting.

DETAILED DESCRIPTION:
Participants will continue study treatment until disease progression, death, unacceptable toxicity, participant request to stop treatment, investigator decision or study termination by the sponsor.

Not all substudies may be active and/or open to enrollment at a given time. Not all study centers may be participating in every substudy. MBC substudy will be the first to enroll - thus the information reflected in the enrollment number, arms/interventions, outcome measures, and eligibility criteria only include MBC at this time.

ELIGIBILITY:
Inclusion Criteria (all substudies):

* Participants must have at least one measurable lesion as defined by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) must be 0 to 1.
* Life expectancy of at least 3 months
* Participants must have recovered from all AEs due to previous therapies, procedures, and surgeries to baseline severity or ≤Grade 1 per NCI CTCAE v5.0 except for AEs not deemed reversible which do not constitute a safety risk by Investigator judgment

MBC substudy:

* Histologically confirmed invasive HER2 positive breast cancer
* Available tumor tissue (FFPE slides or block). A fresh biopsy is preferred but optional.
* Received at least one prior line of therapy including T-DXd for locally advanced/metastatic HER2 positive breast cancer. Prior neoadjuvant therapy which resulted in relapse within 6 months of completion of T-DXd will be considered a line of treatment for metastatic disease.
* Progressed on or following the most recent line of therapy
* Eligible to receive one of the following chemotherapy options (capecitabine, eribulin, gemcitabine, paclitaxel or vinorelbine)
* LVEF ≥50%
* Adequate renal function (estimated creatinine clearance ≥30 mL/min as calculated using the Cockroft-Gault equation
* Adequate liver function:
* Total bilirubin ≤1.5 x upper limit of normal (ULN) (≤3.0 x ULN if the participant has documented Gilbert syndrome);
* Aspartate and alanine transaminase (AST and ALT) ≤3 x ULN (≤5.0 x ULN if liver involved by metastatic disease).

Exclusion Criteria (all substudies):

* Participants with known CNS metastases unless treated and stable prior to enrollment
* Following anti-cancer therapy with insufficient washout before C1D1:

  1. chemotherapy, hormonal therapy, radiation therapy or small molecule anti-cancer therapy within 14 days or 5 half-lives (whichever is shorter) of C1D1.
  2. Immune therapy or other biologic therapy (e.g., monoclonal antibodies, antibody-drug conjugates) for the treatment of cancer for: 28 days or 5 half-lives (whichever is shorter) of C1D1)
* Prior exposure to any anti-CD47 or anti-SIRPα agent.
* History of autoimmune hemolytic anemia, autoimmune thrombocytopenia, or hemolytic transfusion reaction.
* Had an allogeneic tissue/solid organ transplant.
* Any active, unstable cardiovascular disease
* Intolerance to or who have had a severe allergic or anaphylactic reaction to antibodies or infused therapeutic proteins or participants who have had a severe allergic or anaphylactic reaction to any of the substances included in the study drug (including excipients).
* Has an active autoimmune disease that has required systemic treatment in past 2 years

MBC substudy:

* Has a diagnosis of complete dihydropyrimidine dehydrogenase (DPD) deficiency or significant toxicity with prior flurouracil (5FU) based regimen
* Other primary malignancy within 2 years
* Any condition that would be contraindicated to receiving trastuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MBC substudy: Overall Response Rate (ORR) using RECIST v1.1 based on BICR assessment | Approximately 6 months after the last participant is enrolled
  Evaluate the ORR of evorpacept in combination with trastuzumab and single-agent chemotherapy in the sub-population of participants with metastatic HER2-positive ctDNA-positive breast cancer. ORR is defined as a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) using RECIST v1.1 based on BICR assessment.

SECONDARY OUTCOMES:
MBC substudy: Overall Response Rate (ORR) based on Investigator assessment | Approximately 6 months after the last participant is enrolled
  Evaluate the ORR of evorpacept in combination with trastuzumab and single-agent chemotherapy in the sub-population of participants with metastatic HER2-positive ctDNA-positive breast cancer by levels of CD47 expression. ORR is defined as a best overall response (BOR) of confirmed complete response (CR) or partial response (PR) based on Investigator Assessment.
MBC substudy: Clinical Benefit Rate (CBR) using RECIST v1.1 based on BICR and Investigator assessment | Approximately 6 months after the last participant is enrolled
  Evaluate the CBR of evorpacept in combination with trastuzumab and single-agent chemotherapy in the sub-population of participants with metastatic HER2-positive ctDNA-positive breast cancer. CBR is defined as the proportion of participants whose BOR is confirmed PR, confirmed CR, or SD with duration >6 months using RECIST v1.1 based on BICR and Investigator assessment.
MBC substudy: Duration of Response (DoR) using RECIST v1.1 based on BICR and Investigator assessment | Approximately 6 months after the last participant is enrolled
  Evaluate the DoR of evorpacept in combination with trastuzumab and single-agent chemotherapy in the sub-population of participants with metastatic HER2-positive ctDNA-positive breast cancer. DoR is measured from the time measurement criteria are first met for CR / PR (whichever is first recorded) until documented progressive disease or death from any cause, whichever occurs first using RECIST v1.1 based on BICR and Investigator assessment.
MBC substudy: Progression-Free Survival (PFS) using RECIST v1.1 based on BICR and Investigator assessment | Approximately 6 months after the last participant is enrolled
  Evaluate the PFS of evorpacept in combination with trastuzumab and single-agent chemotherapy in the sub-population of participants with metastatic HER2-positive ctDNA-positive breast cancer. PFS is measured from the date of enrollment until documented progressive disease or death from any cause, whichever occurs first, using RECIST v1.1 based on BICR and Investigator assessment
MBC substudy: Overall Survival (OS) | Approximately 6 months after the last participant is enrolled
  Evaluate the OS of evorpacept in combination with trastuzumab and single-agent chemotherapy in the sub-population of participants with metastatic HER2-positive ctDNA-positive breast cancer. OS is defined as the time from the date of enrollment until death.
MBC substudy: Number of participants with adverse events (AEs) and with laboratory abnormalities | Enrollment to 28 days after the last administration of the study drug
  AEs as characterized by type, frequency, severity (as graded by NCI CTCAE v5.0), timing, seriousness, and relationship to study drug. Laboratory abnormalities as characterized by type, frequency, severity, and timing.
All substudies: Maximum Concentration (Cmax) | Approximately 6 months after the last participant is enrolled
  To evaluate the Cmax of evorpacept
All substudies: Time at Maximum Concentration (Tmax) | Approximately 6 months after the last participant is enrolled
  To evaluate the Tmax of evorpacept
All substudies: Area under the Concentration-Time Curve (AUC) | Approximately 6 months after the last participant is enrolled
  To evaluate the AUC of evorpacept
All substudies: Clearance (CL) | Approximately 6 months after the last participant is enrolled
  To evaluate the CL of evorpacept
All substudies: Terminal elimination half-life (t1/2) | Approximately 6 months after the last participant is enrolled
  To evaluate the t1/2 of evorpacept
All substudies: Evaluate the immunogenicity of evorpacept | Approximately 6 months after the last participant is enrolled
  Measured by presence of human serum ADA (anti-evorpacept antibodies)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - Saint Mary's Regional Hospital - Cancer Centers of Colorado, Grand Junction, Colorado
  - The George Washington Medical facility Associates, Washington D.C., District of Columbia
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - HealthPartners Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Oncology Hematology West, Pc Dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Gabrail Cancer Center, Canton, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No